CLINICAL TRIAL: NCT01234883
Title: A Double-Blind, Randomized, Comparative Efficacy and Safety Trial of Intravenous Solutions for the Treatment of Moderate to Severe Dehydration in Children With Acute Gastroenteritis
Brief Title: Intravenous (IV) Solutions for Dehydration in Children With Gastroenteritis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSPIVTUSA001
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-03

CONDITIONS: Dehydration; Gastroenteritis
Keywords: dehydration; gastroenteritis
MeSH Terms: conditions — Dehydration; Gastroenteritis | interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- multiple electrolyte solution (Experimental): Subjects were randomized to receive either multiple electrolyte solution or saline. These solutions were administered IV at 10-20 mL/kg until the subject appeared clinically rehydrated as assessed by the clinician. The selected dose for these solutions is considered standard of care when treating clinical dehydration in children and is consistent with product labeling.
  Interventions: Drug: multiple electrolyte solution
- saline (Active Comparator): Subjects were randomized to receive either multiple electrolyte solution or saline. These solutions were administered IV at 10-20 mL/kg until the subject appeared clinically rehydrated as assessed by the clinician. The selected dose for these solutions is considered standard of care when treating clinical dehydration in children and is consistent with product labeling.
  Interventions: Drug: saline

INTERVENTIONS:
Drug: multiple electrolyte solution — IV multiple electrolyte solution dosed as clinically indicated for rehydration
  Other Names: Plasma Lyte A Injection pH 7.4 (Multiple Electrolytes Injection, Type 1, USP)
  Arms: multiple electrolyte solution
Drug: saline — IV solutions dosed as clinically indicated for rehydration
  Other Names: 0.9% Normal Saline
  Arms: saline

SUMMARY:
The primary objective of this study is to compare the efficacy and safety of the use of a multiple electrolyte solution to the use of saline for the treatment of moderate to severe dehydration due to acute gastroenteritis (AGE) in children.

DETAILED DESCRIPTION:
The primary objective of this study was to compare the efficacy and safety of the use of Plasma Lyte A to the use of NS for the treatment of moderate to severe dehydration and amelioration of metabolic acidosis due to AGE in children (≥ 6 months to < 11 years of age) by measuring serum bicarbonate levels.

ELIGIBILITY:
Inclusion Criteria:

1. AGE (etiology: viral or other) resulting in presentation to the ED deemed in need of IV rehydration. In the 24 hours prior to presentation, the subject experienced at least 3 episodes of diarrhea (loose and/or watery stools) and/or nonbilious vomiting.
2. Moderate to severe dehydration (as assessed by Gorelick score13 ≥ 4
3. ≥ 6 months to < 11 years of age.
4. Healthy except for the underlying etiology of AGE.
5. Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved written ICFs and privacy language per national regulations (eg, Health Insurance Portability and Accountability Act [HIPAA], Personal Information Protection and Electronic Documents Act [PIPEDA]) were obtained from the parent/guardian prior to any study-related procedures.

Exclusion Criteria:

1. AGE that did not require IV rehydration per the clinician.
2. Gorelick score ≤ 3
3. Bilious vomiting.
4. Received > 20 mL/kg IV fluid bolus within the 4 hours prior to study enrollment (ie, Hour -4 to Hour 0).
5. Diarrhea lasting > 7 days prior to presentation to the ED.
6. Chronic vomiting disorder.
7. Grossly bloody diarrhea.
8. Chronic diarrheal disorder.
9. Known hyponatremia (sodium < 130 mmol/L [< 130 mEq/L]) within 72 hours prior to enrollment.
10. Known hypernatremia (sodium > 155 mmol/L [> 155 mEq/L]) within 72 hours prior to enrollment.
11. Known hypokalemia (potassium < 3.0 mmol/L [< 3.0 mEq/L]) within 72 hours prior to enrollment.
12. Known hyperkalemia (potassium > 5.5 mmol/L [> 5.5 mEq/L]) within 72 hours prior to enrollment.
13. The use of prohibited medications:

    * Antacids within 24 hours prior to presentation to the ED and during the study.
    * Anti-diarrhea medication within 24 hours prior to presentation to the ED and during the study.
    * The systemic use of corticosteroids/corticotropins was prohibited within 72 hours of enrollment.
14. Chronic health condition affecting the ability to tolerate fluids or those that result in electrolyte abnormalities (eg, chronic renal, cardiac, or pulmonary diagnoses), or abnormalities of sodium or potassium handling (eg, endocrine disorders, medications).
15. Any reason for urgent or emergency hospital admission or ED stays of > 12 hours within 14 days preceding presentation to the ED.
16. Any medical condition likely to interfere with the subject's ability to fully complete all protocol-specified interventions, the ability to undergo all protocol-specified assessments, or likely to prolong the subject's need for medical attention beyond that required for treatment of dehydration.
17. Participation in a study of any investigational drug or device concomitantly or within 30 days prior to enrollment in this study, including previous enrollment in this study.
18. Subject with a > 50% expected chance of dying within 6 months, in the Investigator's opinion.
19. Known hypersensitivity to either of the investigational products.
20. Other serious acute or active conditions that, in the Investigator's opinion, precluded participation in this study.

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Drew Jones, MD, Study Director — Baxter Healthcare
Locations (9):
- United States (7):
  - Emory University/Children's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Hospital of Atlanta at Scottish Rite, Atlanta, Georgia
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia

REFERENCES:
- [Derived] Allen CH, Goldman RD, Bhatt S, Simon HK, Gorelick MH, Spandorfer PR, Spiro DM, Mace SE, Johnson DW, Higginbotham EA, Du H, Smyth BJ, Schermer CR, Goldstein SL. A randomized trial of Plasma-Lyte A and 0.9 % sodium chloride in acute pediatric gastroenteritis. BMC Pediatr. 2016 Aug 2;16:117. doi: 10.1186/s12887-016-0652-4. PMID 27480410

RESULTS

PARTICIPANT FLOW:
Groups:
- Multiple Electrolyte Solution: Plasma Lyte A Injection pH 7.4 (Multiple Electrolytes Injection, Type 1, USP): IV multiple electrolyte solution dosed as clinically indicated for rehydration.
- Saline: 0.9% Normal Saline: IV saline solution dosed as clinically indicated for rehydration
Period: Overall Study
Arm/Group | Multiple Electrolyte Solution | Saline
Started | 51 | 49
Completed | 41 | 36
Not Completed | 10 | 13
Not completed — Early treatment release | 8 | 10
Not completed — Parent/guardian withdrew consent | 1 | 2
Not completed — Technical difficulties with IV infusion | 0 | 1
Not completed — Inclusion/exclusion failure | 1 | 0

BASELINE CHARACTERISTICS:
Population: The ITT population was all subjects who were randomized to receive study treatment. Baseline characteristics include data from participants in the ITT population.
Groups:
- Plasma-Lyte A: multiple electrolyte solution: IV multiple electrolyte solution dosed as clinically indicated for rehydration
- 0.9% Saline: saline: IV saline solution dosed as clinically indicated for rehydration
- Total: Total of all reporting groups
Arm/Group | Plasma-Lyte A | 0.9% Saline | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Continuous [Mean (Standard Deviation); unit: months] | 55.22 (32.84) [.5 to 11] | 38.14 (31.35) [.5 to <11] | 46.85 (33.09) [.5 to 11]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 18 | 45
  Male | 24 | 31 | 55

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Venous Serum Bicarbonate at 4 Hours From Start of Intravenous (IV)
Description: The primary efficacy variable was venous serum bicarbonate (marker of metabolic acidosis) at Hour 4 (+/- 1 hour) from the start of the First IV Bolus.
Time Frame: Day 1 (4 Hours after start of IV)
Population: The mITT population is all subjects with Baseline bicarbonate value ≤ 22 mmol/L. The mITT population was used for efficacy evaluation. The AT analysis set was defined as all subjects who received at least 5 mL of study treatment and were classified according to actual treatment received. AT population was used for AE analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Saline: saline: IV saline solution dosed as clinically indicated for rehydration
Arm/Group | Multiple Electrolyte Solution | Saline
Number analyzed (Participants) | 39 | 38
mmol/L | 1.63 (2.54) | 0.00 (2.25)
Statistical Analysis 1: Comparison: Multiple Electrolyte Solution vs Saline; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Description: Treatment emergent SAE and AEs reported on As Treated Population; events starting after the onset of study treatment administration through end of the safety follow-up period.
Arm/Group | Multiple Electrolyte Solution | Saline
Serious Adverse Events (participants affected / at risk) | 1/46 | 0/45
Other Adverse Events (participants affected / at risk) | 13/46 | 8/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multiple Electrolyte Solution (N=46) | Saline (N=45)
Pancreatic enzyme increase (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multiple Electrolyte Solution (N=46) | Saline (N=45)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0)
Injection site extravasation (General disorders) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 2 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Pancreatic Enzymes Increased (Investigations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination of study due to low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other